CLINICAL TRIAL: NCT00138593
Title: Extension to a Study of the Efficacy and Safety of Vildagliptin in Patients With Type 2 Diabetes With HbA1c 9-11%
Brief Title: Extension to a Study of the Efficacy and Safety of Vildagliptin in Patients With Type 2 Diabetes With Hemoglobin A1c (HbA1c) 9-11%
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLAF237A2329E1
Record Dates: First submitted 2005-08-27; First posted 2005-08-30 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 diabetes; vildagliptin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin

INTERVENTIONS:
Drug: vildagliptin

SUMMARY:
This study is not being conducted in the United States. This is a 52-week extension to a study to assess the safety and effectiveness of two doses of vildagliptin, an unapproved drug, in lowering overall blood glucose levels in people with type 2 diabetes who had not previously been treated with drug therapy to lower their blood sugar and whose blood sugar levels were in a specified range. The purpose of the extension study is to gather data on the long term safety and effectiveness of vildagliptin in people with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Only patients successfully completing study CLAF237A2329 are eligible
* Written informed consent
* HbA1c reduction from baseline to week 12 (visit 5) of the core study is greater than or equal to 0.3 absolute units
* Ability to comply with all study requirements

Exclusion Criteria:

* Premature discontinuation from study CLAF237A2329
* Other protocol-defined exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180
Dates: Start 2004-07; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Safety in combination with pioglitizone after 52 weeks of treatment
Change from baseline in HbA1c at 52 weeks

SECONDARY OUTCOMES:
Change from baseline in fasting plasma glucose at 52 weeks
Change from baseline in fasting lipids at 52 weeks
Change from baseline in body weight at 52 weeks
Change from baseline in HOMA B at 52 weeks
Change from baseline in HOMA IR at 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Pharmaceuticals, Basel, Switzerland

REFERENCES:
- [Result] Ligueros-Saylan M, Foley JE, Schweizer A, Couturier A, Kothny W. An assessment of adverse effects of vildagliptin versus comparators on the liver, the pancreas, the immune system, the skin and in patients with impaired renal function from a large pooled database of Phase II and III clinical trials. Diabetes Obes Metab. 2010 Jun;12(6):495-509. doi: 10.1111/j.1463-1326.2010.01214.x. PMID 20518805